CLINICAL TRIAL: NCT01142947
Title: Study of Asthma Phenotypes and Pharmacogenomic Interactions by Race-Ethnicity (SAPPHIRE)
Acronym: SAPPHIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, keoki williams, Senior Scientist, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AI079139
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Asthma
Keywords: Inhaled corticosteroids; Asthma; Pharmacogenomics; Genome wide association study; Admixture mapping; Continental population groups
MeSH Terms: conditions — Asthma | interventions — Beclomethasone

STUDY DESIGN:
Intervention Model Description: Discovery set for ICS treatment response biomarker analysis
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- beclomethasone dipropionate (BD) (Other): Patients who meet eligibility criteria will be treated with 6 weeks of beclomethasone dipropionate to assess change in pulmonary function and asthma control. These change will be used as phenotypes in a genetic association study. There is no placebo group.
  Interventions: Drug: beclomethasone dipropionate

INTERVENTIONS:
Drug: beclomethasone dipropionate — 160 mcg twice a day (320 mcg per day total)

SUMMARY:
Inhaled corticosteroids (ICS) are considered first-line treatment for persistent asthma, yet little is known about the genetic factors that influence response to this therapy. This study seeks to quantify response to ICS therapy in African American and white patients, as well as look for genetic markers that predict treatment response.

DETAILED DESCRIPTION:
Inhaled corticosteroids (ICS) are considered first-line therapy for the management and control of patients with persistent asthma. Use of inhaled steroids has been associated with improved lung function, diminished symptoms, and fewer exacerbations. However studies show considerable inter-subject variability in ICS response. It has also been estimated that corticosteroid resistance accounts for half of all asthma-related health care costs. Therefore, identifying factors associated with ICS response is both clinical and economically important. African-American patients have been understudied with respect to genetic predictors of asthma controller medication response, and to date there have been no sufficiently powered genome-wide association studies of ICS treatment response among African American individuals with asthma. This issue is of particular importance, since African-American individuals are disproportionately affected by asthma-related complications. In this proposal, we seek to identify novel genetic loci associated with ICS treatment responsiveness (defined by the change in Asthma Control Test score) among African American individuals treated with beclomethasone dipropionate (BD) for 6 weeks. We will attempt to validate loci identified in the discovery set by 1) reassessing these variants for their interaction with ICS treatment on asthma exacerbations in a separate group of African American individuals with asthma, and 2) by reexamining the genetic association with change in asthma control among similarly treated (i.e., treatment with 6 weeks of BD) European Americans with asthma.

ELIGIBILITY:
Inclusion Criteria for Discovery Group:

* Age 12-56 years
* Physician diagnosis of asthma (identified by using encounter data prior to screening and by the survey administered at the clinic visit)
* Bronchodilator reversibility on pulmonary function testing (i.e., improvement in baseline FEV1 of >12%)
* African-American/Black self-reported race-ethnicity

Exclusion Criteria for Discovery Group:

* Smoking in the preceding year or <10 pack-year smoking history total
* Pregnant at the time of enrollment or intending to get pregnant during the 6-week treatment period
* Oral or inhaled corticosteroid use in the 4 weeks preceding enrollment
* Prior diagnosis of chronic obstructive pulmonary disease or emphysema
* Prior diagnosis of congestive heart failure
* Self-reported race not African-American/Black or Hispanic ethnicity (these groups could be included in Replication/Validation group)

Ages: 12 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 362 (Actual)
Dates: Start 2007-10; Primary Completion 2017-02 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Keoki Williams, MD, MPH, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Levin AM, Gui H, Hernandez-Pacheco N, Yang M, Xiao S, Yang JJ, Hochstadt S, Barczak AJ, Eckalbar WL, Rynkowski D, Samedy LA, Kwok PY, Pino-Yanes M, Erle DJ, Lanfear DE, Burchard EG, Williams LK. Integrative approach identifies corticosteroid response variant in diverse populations with asthma. J Allergy Clin Immunol. 2019 May;143(5):1791-1802. doi: 10.1016/j.jaci.2018.09.034. Epub 2018 Oct 24. PMID 30367910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 362 self-reported African American enrolled in 6-week treatment with inhaled beclomethasone dipropionate; 291 returned at the end of treatment; 262 with measurable medication adherence; 244 with genome-wide genotype data.
Groups:
- Beclomethasone Dipropionate (BD): Patients who meet eligibility criteria will be treated with 6 weeks of beclomethasone dipropionate to assess change in asthma control. This change will be the phenotype used in discovery for the genetic association study. There is no placebo group.
  beclomethasone dipropionate: 160 mcg twice a day (320 mcg per day total)
Period: Overall Study
Arm/Group | Beclomethasone Dipropionate (BD)
Started | 362
Completed | 244
Not Completed | 118

BASELINE CHARACTERISTICS:
Arm/Group | Beclomethasone Dipropionate (BD)
Number analyzed (Participants) | 362
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216
  Male | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 362
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Proportion of African Genetic Ancestry [Mean (Standard Deviation); unit: % African Ancestry (within individuals)] — Population: Some individuals did not have the genome wide genotype data needed to assess genetic ancestry.
  % African Ancestry (within individuals)
    number analyzed (Participants) | 330
    (all) | 80.6 (8.7)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meters squared] | 32.4 (9.5)
Smoking Status [Count of Participants; unit: Participants] — Population: Smoking status missing on seven individuals
  Participants
    number analyzed (Participants) | 355
    Never Smoker | 315
    Past Smoker | 37
    Current Smoker | 3
Initial Asthma Control Test Score [Mean (Standard Deviation); unit: Composite Score] — The Asthma Control Test comprises five questions, each with a Likert Scale of 1 to 5. Therefore, the composite score for an individual ranges from 5 to 25. Higher composite scores denote better controlled asthma. Population: Initial ACT score missing in 8 individuals
  Composite Score
    number analyzed (Participants) | 354
    (all) | 17.8 (5.0)
Percent of Predicted Forced Expiratory Volume at 1 Second [Mean (Standard Deviation); unit: % of the predicted FEV1] — The predicted forced expiratory volume at one second (FEV1) is derived from predictive equations derived from population based studies (Hankinson et al. Am J Respir Crit Care Med. 1999 Jan;159(1):179-87.). The percent of predicted for an individual is derived by dividing the measured FEV1 for that individual by their predicted measure (the later is based on an individual's age, sex, and race-ethnicity).
  % of the predicted FEV1 | 73.0 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Control Test Score
Description: Patients will be treated with 6 weeks of inhaled beclomethasone diproprionate (BD) treatment and the change in Asthma Control Test (ACT) quantified. The composite ACT score measured at each time point ranged from 5-25 (with higher scores reflective of better asthma control). Therefore, the absolute change in ACT score from before to after treatment could range from -20 to +20.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: change in composite score
Arm/Group | Beclomethasone Dipropionate (BD)
Number analyzed (Participants) | 244
change in composite score | 3.32 (4.47)

ADVERSE EVENTS:
Time Frame: 6 weeks of treatment with inhaled beclomethasone dipropionate.
Arm/Group | Beclomethasone Dipropionate (BD)
All-Cause Mortality (participants affected / at risk) | 0/362
Serious Adverse Events (participants affected / at risk) | 0/362
Other Adverse Events (participants affected / at risk) | 0/362

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT01142947/Prot_SAP_000.pdf